CLINICAL TRIAL: NCT06876168
Title: Virtual Reality in ICU (PARTNER) - A Research Study About Engaging in Strategies to Promote Relaxation, Improve Your Mood, and Stimulate Thinking in the Intensive Care Setting
Brief Title: Virtual Reality in ICU - PARTNER
Acronym: VR-PARTNER
Status: Recruiting | Type: Observational
Sponsor: Kirby Mayer (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Kirby Mayer, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 97957; R43AT013038 (NIH)
Record Dates: First submitted 2025-02-24; First posted 2025-03-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure; Sepsis
Keywords: virtual reality; intensive care unit; sepsis; acute respiratory failure
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- VR-PARTNER: Participants in ICU

SUMMARY:
This project is designed to have patients participate in a virtual environment with various tasks such as breathing exercises, games to help the brain, and techniques that promote relaxation while hospitalized in the Intensive Care Unit (ICU). The participation in research will last about 5 days and take about 15 to 45 minutes each day.

DETAILED DESCRIPTION:
This is a research study about interacting and engaging in strategies to promote relaxation, improve mood, and stimulate thinking in patients in the Intensive Care Unit (ICU) in the hospital; called PARTNER. PARTNER is played by using a readily available Virtual Reality headset while patients are in the ICU. The researchers hope to learn if engaging with exercises for emotional health and cognitive function reduces delirium and loneliness in the hospital. If patients agree, the patients will be asked to play PARNTER, with a Virtual Reality (VR) device to connect them to a virtual environment with games and/or relaxing scenes while in the ICU. The Virtual environment may include things such as breathing exercise, mindfulness training, and relaxation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to ICU at University of Kentucky for acute respiratory failure, sepsis or other

Exclusion Criteria:

* Are less than 18 years of age
* Have a pre-existing neurologic disorder
* Have a pre-existing emotional or personality disorder
* Have a history or active mental health disorder or disease
* Experienced an acute neurologic event (e.g., stroke)
* Are currently pregnant
* Are a prisoner
* Receiving hospice care
* Have existing open wounds or pressure ulcers on head or neck

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit at University of Kentucky with sepsis or acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | From enrollment to end of treatment (5 sessions); Day 1 through Day 5
  System Usability Scale - describing the ease of use of the procedure and device
Completion rate - feasibility | From enrollment to the end of treatment (5 sessions); Day 1 through Day 5
  Feasibility will be defined as the number of sessions completed as compared to the number of days after extubation (or BiPap removal, HFNC removal) and discharge from ICU/hospital.

SECONDARY OUTCOMES:
MoCA | Through study completion, typically occurring at hospital discharge or within 10 days of hospital discharge
  Montreal Cognitive Assessment. The Montreal Cognitive Assessment (MoCA) is screening tool for detecting mild cognitive impairment (MCI) and early signs of dementia. It assesses various cognitive domains, including attention, memory, language, visuospatial skills, and executive function.The MoCA Scoring Range:
  Total Score: 0 to 30, Normal Cognition: 26-30, Mild Cognitive Impairment (MCI): 18-25, Moderate Cognitive Impairment: 10-17, Severe Cognitive Impairment: <10. A score below 26 generally indicates cognitive impairment, though adjustments may be made for education level (e.g., adding 1 point for individuals with ≤12 years of education). Researchers are trained and certified to give the assessment.
Hospital Anxiety and Depression Survey (HADS) | Through study completion, occurring at the time of hospital discharge, or at a 10, 30, or 60-day post-hospital discharge follow-up, conducted either at the ICU Recovery Clinic or by telephone.
  Hospital Anxiety and Depression is an instrument that measures anxiety and depression. The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire designed to assess anxiety and depression in patients, particularly in hospital and clinical settings. It consists of 14 items, divided into two subscales: HADS-A (Anxiety): 7 items HADS-D (Depression): 7 items; Each item is scored from 0 to 3, with a total possible score of 0 to 21 for each subscale. HADS Scoring Range: 0-7: Normal; 8-10: Borderline case (mild symptoms); 11-21: Clinical case (moderate to severe symptoms).
IES-R | Through study completion, occurring at the time of hospital discharge, or at a 10, 30, or 60-day post-hospital discharge follow-up, conducted either at the ICU Recovery Clinic or by telephone.
  Impact of Events Scale - Revised (IES_R). The Impact of Event Scale - Revised (IES-R) is a self-report measure used to assess psychological distress and symptoms of post-traumatic stress disorder (PTSD) following a traumatic event. It consists of 22 items, divided into three symptom clusters: 1) Intrusion (8 items) - recurrent thoughts, nightmares, flashbacks; 2) Avoidance (8 items) - emotional numbness, avoiding reminders; 3) Hyperarousal (6 items) - irritability, hypervigilance, difficulty sleeping. The IES-R Scoring Range has a Total Score Range of 0-88 with: 0-23: Minimal impact, 24-32: Mild impact (possible PTSD concern), 33-36: Moderate impact (likely PTSD), ≥37: Severe impact (PTSD highly probable). Higher scores indicate greater distress and a higher likelihood of PTSD. The IES-R is not a diagnostic tool but helps assess symptom severity.
EQ5D | Through study completion, typically occurring at hospital discharge or within 10 days of hospital discharge
  The EQ-5D is a standardized, self-reported health-related quality of life (HRQoL) measure developed by the EuroQol Group. It assesses five dimensions of health: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Each dimension is rated on a 5-level (EQ-5D-5L) scale.It also includes a visual analog scale (EQ-VAS), where patients rate their overall health on a 0-100 scale (0 = worst health, 100 = best health).

CONTACTS AND LOCATIONS:
Overall Officials: Kirby P. Mayer, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.